CLINICAL TRIAL: NCT06597981
Title: Development and Testing of a Dyadic Empowerment-based Sport Stacking Program to Improve Health Outcomes of People With Mild Dementia and Their Family Caregivers
Brief Title: Dyadic Sport Stacking Program for Mild Dementia and Their Family Caregivers
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Yang Ziying, Principal Investigator, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UW 24-395
Record Dates: First submitted 2024-09-12; First posted 2024-09-19 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-09

CONDITIONS: Dementia; Family Caregivers; Dyadic Intervention; Health Related Quality of Life; Cognition
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dyadic empowerment-based sport stacking group (Experimental)
  Interventions: Behavioral: Dyadic empowerment-based sport stacking
- Basic education group (Active Comparator)
  Interventions: Other: Basic education

INTERVENTIONS:
Behavioral: Dyadic empowerment-based sport stacking — For the intervention group, the care dyads will receive an 18-week dyadic empowerment-based sport stacking program, which is divided into two phases: the active phase (weeks 1-12) and the maintenance phase (weeks 13-18). In the active phase, the care dyads will engage in three online sessions in small groups (3-5 dyads/group) and three check-up/support sessions. Three online sessions will be scheduled at weeks 1, 3, and 9 during the 12-week active phase. They will also be required to engage in self-practice at home for at least 30 minutes per day, five times per week during this time according to their training schedule. In the maintenance phase, there will be three online sessions in small groups (3-5 dyads/group). Three online sessions will be scheduled at weeks 13, 16, and 18. The dyads will continue their self-practice at home (at least 30 minutes/day, five times/week) for 6 weeks.
  Arms: Dyadic empowerment-based sport stacking group
Other: Basic education — Participants in the control group will receive basic education on dementia caregiving, which will comprise three group-based (3-5 dyads/group) online meetings in the same schedule as the intervention group (1st, 3rd, 9th week).
  Arms: Basic education group

SUMMARY:
The goal of this clinical trial is to develop and test a dyadic empowerment-based sport stacking program to improve health outcomes of people with mild dementia and their family caregivers.

The research hypotheses to be tested are:

i) People with dementia who receive the dyadic empowerment-based sport stacking program will report a greater improvement in cognitive function, a greater reduction in cognitive and neuropsychiatric symptoms, a greater reduction in depressive symptoms, and a greater improvement in health-related quality of life (HRQOL) at T1 (12th week) and T2 (18th week), compared to the usual care group; ii) Caregivers who receive the dyadic empowerment-based sport stacking program will report less stressful in managing the cognitive and neuropsychiatric symptoms, a greater reduction in depressive symptoms and a greater improvement in HRQOL at T1 (12th week) and T2 (18th week), compared to the usual care group; iii) The care dyads who receive the dyadic empowerment-based sport stacking program will report less dyadic relationship strain at T1 (12th week) and T2 (18th week), compared to the usual care group.

For the intervention group, the care dyads will receive an 18-week dyadic empowerment-based sport stacking program, which is divided into two phases: the active phase (weeks 1-12) and the maintenance phase (weeks 13-18). In the active phase, the care dyads will engage in three online sessions in small groups (3-5 dyads/group) and three check-up/support sessions. Three online sessions will be scheduled at weeks 1, 3, and 9 during the 12-week active phase. They will also be required to engage in self-practice at home for at least 30 minutes per day, five times per week during this time according to their training schedule. In the maintenance phase, there will be three online sessions in small groups (3-5 dyads/group). Three online sessions will be scheduled at weeks 13, 16, and 18. The dyads will continue their self-practice at home (at least 30 minutes/day, five times/week) for 6 weeks.

Participants in the control group will receive basic education on dementia caregiving, which will comprise three group-based (3-5 dyads/group) online meetings in the same schedule as the intervention group (1st, 3rd, 9th week).

ELIGIBILITY:
Inclusion Criteria:

- People living with dementia (PLwD) : i) Clinical diagnosis of dementia, in accordance with the Diagnostic and Statistical Manual of Mental Disorders, fifth edition(DSM-V); ii) a minimum age of 60 years; iii) Clinical Dementia Rating (CDR) score of 1; iv) home-dwelling; v) able to communicate with the research personnel to understand training program and assessments; vi) have adequate hearing and visual function to enable skill learning; vii) informed consent.

- Family caregivers: i) aged 18 years or above; ii) living with or providing care to PLwD at least 4 hours/day; iii) able to understand and communicate in Chinese; iv) have access to smartphone/iPad/laptop and are users of one of these devices; v) consent to participate.

Exclusion Criteria:

- People living with dementia (PLwD) : i) severe mental and behavioral disorders; ii) any acute medical condition precluding participation in the program (e.g., pneumonia and cardiac insufficiency); iii) concurrent participation in other studies.

- Family caregivers: i) physically not able to participate in the sport stacking due to physical problems; ii) suffer from acute psychotic condition; iii) unable to support the PLwD in the delivery of sport stacking sessions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2024-09-19 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Health-related quality of life | baseline before randomization (T0), intermediate test at 12 weeks (T1), and post-test at 18 weeks (T2)
  The Short Form 12-item Health Survey-version two (SF-12v2) scale will be used to obtain the patient's health-related quality of life (HRQOL). The sum scores range from 0 to 100, with a higher score representing better HRQOL.
Global cognition | baseline before randomization (T0), intermediate test at 12 weeks (T1), and post-test at 18 weeks (T2)
  The Alzheimer's Disease Assessment Scale-Cognitive Subscale (ADAS-Cog) will be used to evaluate global cognition. The sum scores range from 0 to 70, with a higher score representing poorer cognitive function.
Relationship quality | baseline before randomization (T0), intermediate test at 12 weeks (T1), and post-test at 18 weeks (T2)
  The Dyadic Relationship Scales (Chinese version, DRS), which includes two independent scales (DRS-patient and DRS-caregiver versions) will be used to measure the quality of dyadic relationship between family dyads. The sum scores of DRS-patient range from 0 to 27 and the sum scores of DRS-caregiver range from 0 to 30, with a higher score representing poorer relationship quality.

SECONDARY OUTCOMES:
Memory function | baseline before randomization (T0), intermediate test at 12 weeks (T1), and post-test at 18 weeks (T2)
  The Auditory Verbal Learning Task (AVLT) will be used to assess their memory.
Processing speed and executive function | baseline before randomization (T0), intermediate test at 12 weeks (T1), and post-test at 18 weeks (T2)
  The Trail-Making Test (TMT) will be used to assess cognitive processing speed and executive function.
Behavioral and psychological symptoms of dementia | baseline before randomization (T0), intermediate test at 12 weeks (T1), and post-test at 18 weeks (T2)
  The Neuropsychiatric Inventory (NPI), which was administered to the caregiver, will be utilized to assess the presence and severity of 12 common behavioral and psychological symptoms of dementia. The sum scores range from 0 to 144, with higher scores representing more severe neuropsychiatric behavioral symptoms.
Expressed emotion | baseline before randomization (T0), intermediate test at 12 weeks (T1), and post-test at 18 weeks (T2)
  The 30-item Family Attitude Scale Chinese version (FAS-C) will be used to measure caregivers' expressed emotion. The sum scores range from 0 to 120, with a higher score representing higher levels of expressed emotion.
Burden | baseline before randomization (T0), intermediate test at 12 weeks (T1), and post-test at 18 weeks (T2)
  The 22-item Zarit burden interview (ZBI, Chinese version) will be used to assess caregivers' burden.
Compliance rate in sport stacking | baseline before randomization (T0), intermediate test at 12 weeks (T1), and post-test at 18 weeks (T2)
  Frequency of dyadic practice and total time will be used to evaluate completion status in sport stacking program.

CONTACTS AND LOCATIONS:
Locations (1):
- the First Affiliated Hospital of Chongqing Medical University, Chongqing, China

IPD SHARING:
Plan to Share IPD: Yes
Data obtained through this study may be provided to qualified researchers with academic interest in dementia. The data will be shared until after publication. The data may be shared through a file that requires a password for access. The personal information of participants has already been replaced with a unique case ID to ensure confidentiality and protect their privacy.
Time Frame: Researchers may submit data requests beginning 9 months after article publication, with access available for up to 24 months. Extensions can be considered on a case-by-case basis.
Access Criteria: Qualified researchers conducting independent scientific research can request access to trial IPD. This access will be granted after the review and approval of a research proposal and Statistical Analysis Plan (SAP), along with the execution of a Data Sharing Agreement (DSA).